CLINICAL TRIAL: NCT03940053
Title: The Efficacy of Arginine in Preventing Cancers. A Single Center, Open, Prospective Study
Brief Title: Prevention of Cancer Development and Progression
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zujiang YU (Other)
Responsible Party: Sponsor-Investigator, Zujiang YU, The director of infectious diseases department, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APT-001
Record Dates: First submitted 2019-05-05; First posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Arginine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observation (No Intervention): Subjects only accept the routine treatment for underlying diseases.
- Intervention (Experimental): Based on the routine treatment for underlying diseases, subjects were administrated by arginine.
  Interventions: Drug: Arginine hydrochloride

INTERVENTIONS:
Drug: Arginine hydrochloride — Arginine hydrochloride injection 5g/dose; 40g/d; ivgtt; sustained medication for 24 days; drug withdrawal for 4 days. Treatment is continued until the levels of tumor marker dropped to normal
  Arms: Intervention

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of arginine in preventing cancer development

DETAILED DESCRIPTION:
Cancer is considered to be the leading cause of death among non-infectious diseases and the most important obstacle to increase life expectancy for every country in the 21st century. However, even if various interventions such as embolization chemotherapy, systemic chemotherapy, radiofrequency ablation, and targeted therapy are widely used in clinical practice, the improvement of patients' survival is still limited. Our previous study found that arginine hydrochloride could significantly promote the apoptosis of liver cancer cells, and inhibit the progression of HCC by prompting the urea cycle. Therefore, our research group has carried out this study to evaluate the efficacy of arginine in preventing cancers.

ELIGIBILITY:
Inclusion Criteria:

* 1. Ages 40-75 years 2. 2 ULN of tumor markers (CEA, AFP, ca-125, ca19-9, NSE, HCG and cyfra21-1) 3. No space-occupying lesions were found by the current imaging examination 4. The major organ function is normal that is meeting the following standards: Blood routine examination: (No blood transfusion, no G-CSF and no medication were corrected within 14 days before screening) a.HB≥80g/L； b.ANC≥1.5×109/L；c.PLT≥50×109/L; Biochemical examination: (ALB was not transfused within 14 days before screening) a. ALB ≥29 g/L； b.ALT and AST<5ULN；c. TBIL ≤3ULN；d.creatinine ≤1.5ULN( albumin and bilirubin, two indicators of Child-Pugh liver function class, can only have one for 2 points) 5. For women of childbearing age, the results of serum/urine pregnancy tests must be negative within 7 days before initiation of treatment. All men and women who participate in the study have to take reliable contraceptive measures within the trial and eight weeks after the trial is completed 6. volunteers must signed informed consent.

Exclusion Criteria:

* 1. patients suffering from any malignant tumors in the past (within 5 years) or at the same time; excluding cured basal cell carcinoma and carcinoma in situs of cervix 2. Patients who are undergoing transplantation or have a history of organ transplantation 3. Patients with an allergic history of arginine hydrochloride 4. The blood pressure cannot be reduced to the normal range by the antihypertensive drug treatment in patients with hypertension(systolic pressure>140 mmHg, diastolic pressure>90 mmHg) 5. Patients with myocardial ischemia or myocardial infarction over grade II or a poorly controlled arrhythmia (including QTc interval: men ≥450 ms; women ≥470 ms) 6.Cardiac functional insufficiency of grade III to IV according to NYHA standard; echocardiography: LVEF<50% 7. Patients with severe organ damage and less than 3 years expected survival time 8. Pregnant or lactating women; fertile patients who are unwilling or unable to adopt effective contraceptives 9. Patients with mental sickness or the history of psychotropic drug abuse 10. Patients with severe infection (unable to control the infection effectively) 11. The researchers believe that any other factors unsuitable for entering into the study.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-05-10 (Estimated); Primary Completion 2024-08-10 (Estimated); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
Incidence | 60 months
  the percentage of patients with cancer from start of treatment to follow-up date of last participant cancers Incidence

SECONDARY OUTCOMES:
tumor markers | 60 months
  the levels of tumor markers in every check point
Chinese Quality of Life Questionnaire - EORTC QLQ-C30 score | 60 months
  The overall enjoyment of life